CLINICAL TRIAL: NCT00678509
Title: Phase I/II Study of Multiple-Vaccine Therapy Using Epitope Peptide Restricted to HLA-A*2402 in Treating Patients With Refractory Breast Cancer
Brief Title: Histocompatibility Leukocyte Antigen (HLA)-A*2402 Restricted Peptide Vaccine Therapy in Patients With Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: Tokyo University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Department of Surgery, The Institute of Medical Science, the University of Tokyo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Breast-A24-I, II
Record Dates: First submitted 2008-05-12; First posted 2008-05-15 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-03

CONDITIONS: Breast Cancer
Keywords: HLA-A*2402; Peptide Vaccine; TTK
MeSH Terms: conditions — Breast Neoplasms | interventions — montanide ISA 51

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Biological: TTK peptide mixed with Montanide ISA 51

INTERVENTIONS:
Biological: TTK peptide mixed with Montanide ISA 51 — Patients will be vaccinated twice a week for 8 weeks. On each vaccination day, TTK peptide (1mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection.

SUMMARY:
The purpose of this study is to evaluate the safety and time to progression of HLA-A*2402 restricted epitope peptide TTK emulsified with Montanide ISA 51.

DETAILED DESCRIPTION:
TTK has been identified as cancer specific molecules especially in breast cancer using genome-wide expression profile analysis by cDNA microarray technique. We have determined the HLA-A*2402 restricted epitope peptide derived from this molecule and identified that this peptide significantly induces the effective tumor specific CTL response in vitro and vivo. According to these findings, in this trial, we evaluate the safety, immunological and clinical response of that peptide. Patients will be vaccinated twice a week for 8 weeks. On each vaccination day, TTK-A24-567 peptide (1mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection. Repeated cycles of vaccine will be administered until patients develop progressive disease or unacceptable toxicity, whichever occurs first. In the phase I study, we evaluate the safety and tolerability of this peptide vaccine. In the following phase II study, we evaluate the immunological and clinical response of this vaccine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or recurrent breast cancer
* Resistant against anthracycline-based and taxane-based chemotherapy or difficult to continue the chemotherapy due to intolerable side effect(s)
* Resistant against trastuzumab or difficult to continue it due to intolerable side effect(s) when her-2 is positive
* ECOG performance status 0-2
* Life expectancy > 3 months
* HLA-A*2402
* Laboratory values as follows

  * 2000/mm3<WBC<15000/mm3
  * Platelet count>100000/mm3
  * Bilirubin < 3.0mg/dl
  * Asparate transaminase < 150IU/L
  * Alanine transaminase < 150IU/L
  * Creatinine < 3.0mg/dl
* Able and willing to give valid written informed consent

Exclusion Criteria:

* Pregnancy(woman of childbearing potential:Refusal or inability to use effective means of contraception)
* Breastfeeding
* Active or uncontrolled infection
* Concurrent treatment with steroids or immunosuppressing agent
* Prior chemotherapy,radiation therapy, or immunotherapy within 4 weeks
* Uncontrolled brain and/or intraspinal
* Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
safety (Phase I: toxicities as assessed by NCI CTCAE version3) and efficacy (Phase II: feasibility as evaluated by RECIST) | 2 months

SECONDARY OUTCOMES:
to evaluate immunological responses | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Masaru Shinozaki, MD/PhD, Principal Investigator — Head, Department of Surgery
Locations (1):
- The Institute of Medical Science, the University of Tokyo, Minato-ku, Tokyo, Japan

REFERENCES:
- See also: Research Hospital, the Institute of Medical Science, the University of Tokyo — http://www.transrec.jp/